CLINICAL TRIAL: NCT03364803
Title: Treatment Outcomes for Patients With Cushing's Syndrome: a Prospective Data Collection Study
Brief Title: Collecting Information About Treatment Results for Patients With Cushing's Syndrome
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 17-592
Record Dates: First submitted 2017-12-01; First posted 2017-12-07 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Cushing's Disease; Cushing Syndrome; Cushing Disease
Keywords: Cushing Syndrome; Cushing's Disease; Cushing Disease; 17-592; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Pituitary ACTH Hypersecretion; Cushing Syndrome | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone; Perceived Stress Scale

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Cushing's Syndrome
  Interventions: Other: Cushing's QoL (Quality of Life Questionnaire); Other: Nottingham Health Profile (NHP); Other: Hospital Anxiety and Depression Scale (HADS); Other: Perceived Stress Scale (PSS); Other: Barratt's Impulsivity Scale (BIS); Other: Beck Depression Inventory (BDI); Other: State-Trait Anxiety Inventory (STAI); Other: State Food Craving Questionnaire-State (FCQ-S); Other: Trait Food Craving Questionnaire-Trait (FCQ-T); Other: Visual Analogue Scale (VAS); Other: Sensitivity to Reinforcement of Addictive and other Primary Rewards (STRAP-R) food variant

INTERVENTIONS:
Other: Cushing's QoL (Quality of Life Questionnaire) — Cushing's QoL is a validated disease specific questionnaire consisting of 12 questions on a five-point Likert scale ranging from always to never. The total score ranges from 12 to 60, with a lower score indicating a greater negative impact on health related QoL. This is converted to a 0-100 scale, 0 indicating the worst and 100 indicating the best QoL
Other: Nottingham Health Profile (NHP) — NHP is used in patients to assess general health and quality of life. This assessment consists of 38 yes/no questions that are subdivided into six scales assessing impairments: pain (eight items), energy level (three items), sleep (five items), emotional reactions (nine items), social isolation (five items) and physical mobility (eight items). A higher score indicates more impairment
Other: Hospital Anxiety and Depression Scale (HADS) — HADS consists of 14 items pertaining to anxiety and depression, with each item measured on a four-point scale. Total scores for the anxiety and depression subscales range from 0 to 21. A higher score indicates greater symptomatology
Other: Perceived Stress Scale (PSS) — The PSS predicts both objective biological markers of stress and increased risk of disease in patients with higher stress levels.
Other: Barratt's Impulsivity Scale (BIS) — BDI and BIS in combination have demonstrated that depression and/or binge eating may be mediating factors for the outcome of obesity
Other: Beck Depression Inventory (BDI) — BDI and BIS in combination have demonstrated that depression and/or binge eating may be mediating factors for the outcome of obesity
Other: State-Trait Anxiety Inventory (STAI) — The STAI provides data to help distinguish between anxiety and depression.
Other: State Food Craving Questionnaire-State (FCQ-S) — The FCQ-S consists of 15 items assessing: desire to eat, anticipation of positive reinforcement from eating, anticipation of negative reinforcement (reduction of negative affect) from eating, lack of control over eating, and (physiological) hunger; higher scores reflect stronger food craving. Participants respond, using a Likert-type scale, how much each item is true of them right now.
Other: Trait Food Craving Questionnaire-Trait (FCQ-T) — Trait food craving will be assessed with the Food Craving Questionnaire-Trait (FCQ-T). The FCQ-T consists of 39 items assessing: intentions/plans to eat, anticipation of positive reinforcement from eating, anticipation of negative reinforcement from eating, lack of control over eating, preoccupation with food, (physiological) hunger, emotions preceding or following food cravings or eating, environmental cues that may elicit food cravings, negative emotions including guilt experienced as a consequence of food cravings, and/or indulging such cravings; higher scores again indicate higher trait craving. Individuals are asked to respond, using a Likert-type scale, how much each item is true of them in general.
Other: Visual Analogue Scale (VAS) — A validated visual analogue scale (VAS) questionnaire will be completed in the fasting state. The VAS consists of 100-mm lines with words anchored at each end describing extreme sensations of hunger, prospective consumption ("How much do you think you can eat?"), fullness, and satisfaction, as well as craving (sweet, salty, fatty or savory). Patients will be asked to make a vertical mark across the line corresponding to their feelings. Quantification will performed by measuring the distance from the left end of the line to the mark.
Other: Sensitivity to Reinforcement of Addictive and other Primary Rewards (STRAP-R) food variant — A validated questionnaire that assesses perceived subjective value attributed to expected/hypothetical foods and other primary reinforcers will be administered. This variant of this questionnaire was initially developed by Dr. Goldstein to assess 'liking' and 'wanting' of expected drug rewards for patients with cocaine addiction. The current assessment uses a modified version to assess 'liking' and 'wanting' for food.

SUMMARY:
The purpose of this study is to follow participants with Cushing's syndrome during the course of their routine care and to form a data registry to study long term participant outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 14 or older
* Active or treated overt Cushing's (due to pituitary, ectopic, or adrenal tumor), mild adrenal Cushing's syndrome (MACS), or a silent corticotroph tumor
* The diagnosis of CS or MACS will be made by the PI, based on the below Endocrine Society guidelines, the patient's clinical presentation, and the PI's judgment.

  * Diagnostic criteria for ACTH-dependent Cushing's are according to the Endocrine Society and European Society of Endocrinology guidelines and include: Elevated 24-hour urinary free cortisol (UFC), normal or elevated plasma ACTH, elevated midnight salivary cortisol levels, or classic dexamethasone suppression testing for CD (morning cortisol > 5 ug/dL after 1 mg overnight of classic 2-day low dose test) and a pituitary lesion on MRI (in the case of pituitary Cushing's). If patient does not have any of these results, pathology of ACTH tumor may confirm presence of disease.
  * Diagnostic criterion for MACS is according to the European Society of Endocrinology guidelines: Classic dexamethasone suppression testing for CS (morning cortisol >1.8 µg/dL after 1 mg overnight) and the presence of an adrenal adenoma.
* Silent corticotroph tumors will be defined by surgical pathology demonstrating positivity for ACTH, in the absence of clinical and biochemical features of Cushing's syndrome.
* In lieu of MRI, surgical, or laboratory reports, physician's assessment note including mention of results will also be used as source for eligibility purposes.

Exclusion Criteria:

* Patients with a diagnosis of iatrogenic Cushing's.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, the protocol investigator, or research team at Memorial Sloan-Kettering Cancer Center (MSKCC). If the investigator is a member of the treatment team, s/he will screen their patient's medical records for suitable research study participants and discuss the study and their potential for enrolling in the research study. Potential subjects contacted by their treating physician will be referred to the investigator/research staff of the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-11-28 (Actual); Primary Completion 2026-11-28 (Estimated); Study Completion 2026-11-28 (Estimated)

PRIMARY OUTCOMES:
Collection of data on Cushing's Syndrome participants before and over time after surgical, medication, and/or radiation therapy. | up to 10 years after treatment

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk-Commack (Limited protocol activity), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org